CLINICAL TRIAL: NCT05353283
Title: PrEP Point-of-Care Brief-Intervention for Adherence Among Young Men Who Have Sex With Men
Acronym: PrEP2-BAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MH122286
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Risk Reduction
Keywords: PrEP; Young MSM; POC monitoring; adherence; motivational interviewing; urine test; tenofovir
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): POC adherence testing by a urine tenofovir assay with motivational interviewing counselling
  Interventions: Behavioral: Motivational Interviewing Counselling; Device: Point-of-care Urine Tenofovir Measurement
- Standard of Care (No Intervention): Adherence counselling provided by the participant's PrEP care provider

INTERVENTIONS:
Behavioral: Motivational Interviewing Counselling — Motivational interviewing-based counseling will be provided to the participant based on the results of the urine test
  Arms: Intervention Arm
Device: Point-of-care Urine Tenofovir Measurement — Urine will be collected and the presence or absence of tenofovir will be measured with the point-of-care urine tenofovir test.
  Arms: Intervention Arm

SUMMARY:
Despite advances in HIV prevention, the HIV incidence among young men who have sex with men (YMSM) is increasing, threatening to derail achievement of the United States End the HIV Epidemic goals. Although, pre-exposure prophylaxis (PrEP) is a highly effective HIV prevention method, adherence was sufficiently low to comprise efficacy among a high proportion of YMSM in multiple clinical trials and demonstration projects. In this study, the investigators will leverage a novel urine point-of-care drug-level test for PrEP adherence, to both enhance and target motivational-interviewing-based adherence counseling among YMSM, with the goal of preventing HIV infections among this critically at-risk group.

DETAILED DESCRIPTION:
Young men who have sex with men (YMSM; ages 15-29 years) have rising HIV incidence in the United States. Pre-exposure prophylaxis (PrEP) is a highly effective medication prevent HIV infection, both at the individual and population level. However, in several clinical trials and demonstration projects among YMSM, a majority of participants had adherence to PrEP sufficiently low to compromise efficacy throughout the study. Unfortunately, pill-counts and self-reported adherence have limitations in this population, and therapeutic drug monitoring using previously available methods requires expensive equipment and specialized staff, meaning it cannot be implemented at the point-of-care (POC). The investigators have developed a novel POC test to measure urine drug-levels to PrEP for the first time, providing the opportunity to target and enhance adherence counseling during a routine clinical visit. Substantial knowledge gaps on the correct counseling approach and framing of the drug-level feedback message must be addressed to use this strategy to improve adherence among YMSM. This study will use a mixed methods approach to test the central hypothesis that an intervention leveraging a POC urine bioassay to detect PrEP adherence can both target and enhance adherence counseling. Brief interventions are a motivational interviewing (MI) counseling approach with wide uptake by primary care providers for substance use prevention and medical therapy adherence. PrEP2-BAY proposes a brief intervention be used as the framework for POC drug-level feedback among YMSM using PrEP. This study will test the acceptability, feasibility, and preliminary impact on long-term adherence, measured through hair tenofovir levels, of the brief intervention in a pilot randomized controlled trial among YMSM. This proposed research plan has the goal of optimizing PrEP's impact through a novel adherence support intervention. The findings of this proposal will lead to a R01 application to test a POC bioassay-enhanced adherence brief intervention among YMSM in a multi-city trial, with the goal of reducing the burden of HIV among MSM.

ELIGIBILITY:
Inclusion Criteria:

* Male sex at birth who has sex with men
* Age 18-30 years-old
* Currently receiving tenofovir-based oral PrEP
* Plans to continue taking daily PrEP over the upcoming 3 months

Exclusion Criteria:

* Participant living with HIV
* Age > 30 years

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants indicating satisfied or very satisfied with the intervention | 3 months
  Number of participants reporting to be "satisfied" or "very satisfied" about their overall experience on a five-point Likert scale

SECONDARY OUTCOMES:
Long-term adherence outcomes | 3 months
  Measure change in tenofovir levels in dried blood spots and/or hair from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spinelli, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco/San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in publicly accessible databases once study is complete and study findings disseminated.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 48 months from start of study
Access Criteria: Investigators conducting PrEP research who contact the Principal Investigator

REFERENCES:
- [Background] Stalter RM, Baeten JM, Donnell D, Spinelli MA, Glidden DV, Rodrigues WC, Wang G, Vincent M, Mugo N, Mujugira A, Marzinke M, Hendrix C, Gandhi M; Partners PrEP Study Team. Urine Tenofovir Levels Measured Using a Novel Immunoassay Predict Human Immunodeficiency Virus Protection. Clin Infect Dis. 2021 Feb 1;72(3):486-489. doi: 10.1093/cid/ciaa785. PMID 33527128
- [Background] Spinelli MA, Rodrigues WC, Wang G, Vincent M, Glidden DV, Okochi H, Stalter R, Defechereux P, Deutsch M, Grant RM, Ngure K, Mugo NR, Baeten JM, Gandhi M; Partners PrEP Study Team. Brief Report: High Accuracy of a Real-Time Urine Antibody-Based Tenofovir Point-of-Care Test Compared With Laboratory-Based ELISA in Diverse Populations. J Acquir Immune Defic Syndr. 2020 Jun 1;84(2):149-152. doi: 10.1097/QAI.0000000000002322. PMID 32167963
- [Background] Gandhi M, Wang G, King R, Rodrigues WC, Vincent M, Glidden DV, Cressey TR, Bacchetti P, Spinelli MA, Okochi H, Siriprakaisil O, Klinbuayaem V, Mugo NR, Ngure K, Drain PK, Baeten JM. Development and validation of the first point-of-care assay to objectively monitor adherence to HIV treatment and prevention in real-time in routine settings. AIDS. 2020 Feb 1;34(2):255-260. doi: 10.1097/QAD.0000000000002395. PMID 31634188
- [Background] Spinelli MA, Glidden DV, Rodrigues WC, Wang G, Vincent M, Okochi H, Kuncze K, Mehrotra M, Defechereux P, Buchbinder SP, Grant RM, Gandhi M. Low tenofovir level in urine by a novel immunoassay is associated with seroconversion in a preexposure prophylaxis demonstration project. AIDS. 2019 Apr 1;33(5):867-872. doi: 10.1097/QAD.0000000000002135. PMID 30649051